CLINICAL TRIAL: NCT00077818
Title: A Prospective, Open-label, Randomized, Parallel-group Investigation to Evaluate the Efficacy and Safety of Enoxaparin Versus Unfractionated Heparin in Subjects Who Present to the Emergency Department With Acute Coronary Syndrome
Brief Title: Enoxaparin Versus Unfractionated Heparin in Subjects Who Present to the Emergency Department With Acute Coronary Syndrome (RESCUE)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: XRP4563B_4001
Expanded Access: Available
Record Dates: First submitted 2004-02-12; First posted 2004-02-16 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — enoxaparin sodium

INTERVENTIONS:
Drug: Enoxaparin sodium

SUMMARY:
The purpose of this study is to determine the efficacy and safety of enoxaparin compared to unfractionated heparin (UFH) for patients diagnosed with Acute Coronary Syndrome (ACS) in the emergency department (ED). Efficacy is assessed by using a composite score consisting of 30-day all-cause mortality, non-fatal myocardial infarction (MI) and recurrent angina requiring revascularization.

ELIGIBILITY:
INCLUSION CRITERIA

* Rest angina lasting at least 10 minutes that is highly suggestive of myocardial ischemia and is not explained by trauma or obvious abnormalities on chest x-ray, occurring within 24 hours of randomization;
* TIMI risk score greater than or equal to 4 (a qualitative test for CK-MB or Troponin may be utilized for screening purposes; however, a quantitative test must still be performed.)

EXCLUSION CRITERIA

* Increased bleeding risk as defined by any of the following:

  * Ischemic stroke within the last year
  * Any previous hemorrhagic stroke, intracranial tumor, or intracranial aneurysm
  * Recent (<1 month) trauma or major surgery (including bypass surgery)
  * Active bleeding (other than minor skin abrasions)
* Impaired hemostasis including any one of the following:

  * Known International Normalized Ratio (INR) >1.5
  * Past or present bleeding disorder (including congenital bleeding disorders such as von Willebrand's disease or hemophilia, acquired bleeding disorders, and unexplained clinically significant bleeding disorders)
  * Known or history of thrombocytopenia (platelet count <100,000/mL)
  * History of thrombocytopenia with glycoprotein IIb/IIIa inhibitor therapy, heparin, or enoxaparin
* Angina from a secondary cause such as:

  * severe, uncontrolled hypertension (systolic blood pressure >180 mm Hg despite treatment)
  * anemia
  * valvular disease
  * congenital heart disease
  * hypertrophic cardiomyopathy
  * restrictive or constrictive cardiomyopathy
  * thyrotoxicosis.
* Bundle branch block not known to be old in the context of angina.
* Undergone a percutaneous coronary intervention (PCI) within the past 24 hours.
* A known allergy to heparin, low molecular weight heparin, pork or pork products.
* Any contraindications to treatment with UFH or LMWH.
* A recent (<48 hours) or planned spinal/epidural anesthesia or puncture.
* Thrombolytic therapy within the preceding 24 hours.
* Any other clinically relevant serious diseases, including severe liver disease or renal failure [creatinine clearance <30 mL/min], rendering implementation of the protocol or interpretation of the study results difficult.
* Treatment with other investigational agents or devices within the previous 30 days, planned use of investigational drugs or devices, or has previously enrolled in this trial.
* Inability to comply with the protocol (e.g., has uncooperative attitude, inability to return for follow-up visits).
* Inability to understand the nature, scope, and possible consequences of the study or is otherwise unable to provide informed consent.
* A prosthetic heart valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-06; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
To assess a composite score that considers the occurrence of all-cause mortality, non-fatal MI, or recurrent angina requiring the need for revascularization | up to 30 days (± 2 days) following randomization

SECONDARY OUTCOMES:
Incidence of major hemorrhage | during the index hospitalization
Incidence of minor hemorrhage | during the index hospitalization
Combined incidence of 30-day all-cause mortality and nonfatal MI | at 30 days
The incidence of 30-day all-cause mortality by itself | At 30 days
Total health care utilization | from baseline (initial hospitalization) through the Day 30 follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Luc Sagnard, Study Director — Sanofi